CLINICAL TRIAL: NCT04930861
Title: Phase 1 Clinical Study of Codivir in Outpatients With COVID-19
Brief Title: Study of Codivir in Patients With COVID-19
Acronym: Codivir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Code Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-01-ZM
Record Dates: First submitted 2021-06-16; First posted 2021-06-18 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-11

CONDITIONS: Covid19
Keywords: Corona; Coronavirus; COVID-19; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Hematologic Tests; COVID-19 Nucleic Acid Testing; Electrocardiography; Physical Examination

STUDY DESIGN:
Intervention Model Description: This is an open label study to evaluate the safety and preliminary efficacy of Codivir in 12 mild or moderate COVID-19 patients and onset of symptoms within 72h prior to their inclusion. Treatment will begin in the hospital, participants will be discharged at Day 4 and continue the treatment up to Day 10 at home.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Covidir (Experimental): Patient (adults aged ≥18 years) with mild or moderate COVID-19 and flu-symptoms onset within 72 hours prior to inclusion. Treatment begins at the hospital. On the 4th day, participants who are well will be discharged and continue treatment up to Day 10 at home. All participants will receive Codivir 20 mg SC 2 x daily.
  Interventions: Drug: Covidir injections; Diagnostic Test: One Step Test; Diagnostic Test: IgM and IgG dosage; Diagnostic Test: RT-PCR SARS-CoV-2; Diagnostic Test: Screening blood test; Diagnostic Test: ECG; Diagnostic Test: Medical evaluation; Diagnostic Test: NEWS-2 score; Diagnostic Test: WHO score

INTERVENTIONS:
Drug: Covidir injections — administration of the investigational product CODIVIR at a dose of 20 mg twice a day subcutaneously.
  Other Names: Experimental drug administration
Diagnostic Test: One Step Test — rapid test for the diagnosis of COVID-19 based on the detection of anti-SARS-CoV-2 in the blood.
  Other Names: Covid-19 test
Diagnostic Test: IgM and IgG dosage — blood collection for dosage of Anti SARS-CoV-2 antibodies.
  Other Names: Blood test
Diagnostic Test: RT-PCR SARS-CoV-2 — detection of viral RNA in nasopharyngeal and oropharyngeal samples by the Real Time Protein Chain Reaction technique.
  Other Names: Covid-19 test
Diagnostic Test: Screening blood test — complete blood count, urea, creatinine, uric acid, sodium, potassium, chloride, calcium, glucose, glycated hemoglobin, alkaline phosphatase (FA), alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubins and fractions ( BTF), total proteins and fractions (PTF), lipid profile (total cholesterol, fractions and triglycerides); coagulogram (TP, aPTT); D-dimer; C-reactive protein; HIV, HBV, HCV serology; Ferritin; fibrinogen, Pregnancy test for non-sterile women.
  Other Names: Blood test
Diagnostic Test: ECG — 12-lead electrocardiogram with report.
  Other Names: Electrocardiogram
Diagnostic Test: Medical evaluation — evaluation by the principal investigator or assistant physician with a complete physical examination.
  Other Names: Physical examination
Diagnostic Test: NEWS-2 score — assessment of the participant by the NEWS-2 score.
Diagnostic Test: WHO score — assessment of the participant by the score of the World Health Organization.

SUMMARY:
This is an open-label study to evaluate the safety and preliminary efficacy of Codivir in 12 mild or moderate COVID-19 patients and onset of symptoms within 72h prior to their inclusion. Treatment will begin in the hospital, participants will be discharged at Day 4 and continue the treatment up to Day 10 at home and followed up to day 28.

DETAILED DESCRIPTION:
Eligible participants who agree to participate will be submitted to safety assessments, an RT-PCR and a quick test for COVID-19. Everyone will receive the treatments indicated for their case, except for other investigational medications. Codivir will be administered in addition to these treatments at a dose of 20 mg SC twice daily for 10 days. Participants will remain hospitalized for the first 3 days.

If they have progressed well, they will continue the treatment up to Day 10 at home, receiving a nurse's home visit twice a day to administer Codivir and collect vital signs. Participants will be followed up to Day 28 by telemedicine. A doctor will call them periodically to monitor the clinical evolution, collect adverse events, concomitant medication and instruct the participants. In case of unfavorable evolution, the participants will remain hospitalized receiving the appropriate care. The investigator will decide whether or not the investigational medication will continue, considering the participant's health and well-being.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 60 years;
2. Male or female;
3. SARS-CoV-2 infection indicated by rapid test and confirmed by RT-PCR.
4. Mild or moderate COVID-19:

   * The oxygen saturation in room air >93%;
   * <30 breaths per minute;
5. No signs of hemodynamic decompensation.
6. Absence of pregnancy in women of childbearing age.
7. Able to understand and comply with the requirements of the protocol.
8. Consent to participate

Exclusion Criteria:

1. Participants in need of O2 supplementation by catheter or mask, invasive mechanical ventilation, or vasopressors.
2. Onset of symptoms or rapid test or positive RT-PCR for more than 72 hours of inclusion.
3. Participants in use or expected to use within 24 hours prior to the inclusion of drugs that are under clinical investigation as a therapeutic option for the treatment of COVID-19 (eg hydroxychloroquine, chloroquine, ivermectin, nitazoxanide, among others) during the study period;
4. Body mass index less than 19.9 or greater than 35;
5. Comorbidities such as: other serious infections, active malignancies, autoimmune diseases, liver, kidney or heart failure; another systemic disease and / or laboratory abnormality, which, in the investigator's opinion, prevent the patient from participating in the study;
6. Concomitant HIV, HBV or HCV infection.
7. Pregnancy or lactation;
8. Participation in another clinical trial in the 12 months preceding inclusion;
9. Anti-COVID-19 vaccination at any time;
10. Vaccination for any other infection in the 4 weeks prior to inclusion;
11. Any condition that increases the risk of participating in the study, in the opinion of the investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-08-09 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events related to the investigational product. | 28 days

SECONDARY OUTCOMES:
Clinical evolution according to the score of the World Health Organization between admission and days 10 and 28. | up to 28 days
Clinical evolution according to NEWS2 score between admission and days 10 and 28. | up to 28 days
RT-PCR negative. | up to 28 days
Evolution of IgM & IgG Anti-SARS-CoV-2. | up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Eynat Finkelshtein, Study Director — Code Pharma
Locations (1):
- Hospital Vera Cruz S A (Campinas-SP), Campinas, State of São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No